CLINICAL TRIAL: NCT00277121
Title: Genetic Origin of Lipid Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Lipid Clinic, The National Hospital, Oslo, Norway (Unknown); Research Institute of Internal Medicine, The National Hospital, Oslo, Norway (Unknown); Ullevaal University Hospital (Other); Norwegian Institute of Public Health (Other Government); Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other); CIGENE, Agricultural University of Norway, Aas, Norway (Other)
Other Study IDs: S-03150 (REK); 02/4746 (SHdir); 10163 (NSD)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2006-01-13 (Estimated); Status verified 2006-01

CONDITIONS: Lipid Disorder
Keywords: Lipid disorder; Gene mutation
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Several lipid disorders are without known genetic origin. The scope of this project is to sequence genes superior involved in lipid and carbohydrate metabolism in patients with severe lipid disorders. The resulting mutations will be tested in suitable in vitro systems to detect their part in development of the specific disease.

DETAILED DESCRIPTION:
See "brief summary" above.

ELIGIBILITY:
Inclusion Criteria:

* proven written informed consent prior to recruitment
* male or female
* 18-55 years old
* patients with severe lipid disorders
* fasting plasma cholesterol, triglyceride or glucose, blood pressure or waist circumference/BMI out of normal range

Exclusion Criteria:

-

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Hilde I Nebb, PhD, Study Chair — Department of Nutrition, University of Oslo; Karianne Solaas, PhD, Principal Investigator — Department of Nutrition, University of Oslo; Monica H Carlsen, Principal Investigator — Department of Nutrition, University of Oslo; Leiv Ose, Dr med, Principal Investigator — Lipid Clinic, The National Hospital; Marit S Nenseter, PhD, Principal Investigator — Research Institute of Internal Medicine, The National Hospital; Kirsten Holven, PhD, Principal Investigator — Research Institute of Internal Medicine, The National Hospital; Bente Halvorsen, PhD, Principal Investigator — Research Institute of Internal Medicine, The National Hospital; Serena Tonstad, Dr med, Principal Investigator — Department of Preventive Medicine, Ullevål university hospital; Håkon Gjessing, PhD, Principal Investigator — Norwegian Institute of Public Health; Per Thorsby, Dr med, Principal Investigator — Hormone laboratory, Aker university hospital; Sigbjørn Lien, PhD, Principal Investigator — Agricultural university of Norway; Paul Berg, PhD, Principal Investigator — Agricultural university of Norway; Kjetil Retterstøl, Dr med, Principal Investigator — Lipid Clinic, The National Hospital
Locations (1):
- Department of Nutrition, University of Oslo, Oslo, Norway